CLINICAL TRIAL: NCT02004106
Title: An Open-Label, Multi-Center, Dose-Escalation, Phase I Study With an Expansion Phase, to Evaluate Safety, Pharmacokinetics and Therapeutic Activity of RO6895882, an Immunocytokine, Consisting of a Variant of Interleukin-2 (IL-2v) Targeting Carcinoembryonic Antigen (CEA) Administered Intravenously, in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Efficacy of RO6895882 in Participants With Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28920; 2013-003041-41 (EudraCT Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (3):
- Part 1: RO6895882 Single Ascending Dose (Experimental): Participants will receive RO6895882 at ascending doses (</= 6 mg) as a single intravenous (IV) infusion.
  Interventions: Drug: RO6895882
- Part 2: RO6895882 Dose Escalation Monotherapy (Experimental): Participants in different cohorts will receive RO6895882 at ascending doses as IV infusion qw, q2w or q3w. After completion of Part 2 all participants have the option to receive the recommended RO6895882 dose once defined in Part 2 at the discretion of investigator.
  Interventions: Drug: RO6895882
- Part 3: RO6895882 MTD Expansion (Experimental): Participants will receive RO6895882 at MTD determined in Part 2 as IV infusion qw, q2w or q3w.
  Interventions: Drug: RO6895882

INTERVENTIONS:
Drug: RO6895882 — Participants will receive RO6895882 at different dose levels and schedules defined in respective arms as IV infusion.

SUMMARY:
This open-label, multi-center, dose-escalation study will evaluate the safety, pharmacokinetics, and therapeutic activity of RO6895882 in participants with Carcinoembryonic Antigen (CEA)-positive solid tumors who have progressed on the standard of care therapy. The study will be conducted in 3 parts. Part 1 will be a single ascending dose study in single participant cohort at low RO6895882 dose (less than or equal to [</=] 6 milligrams [mg]). Part 2 will be a dose-escalation study of RO6895882 monotherapy given every week (qw), every 2 weeks (q2w), and possibly every 3 weeks (q3w). Part 3 will be an expansion phase of the qw, q2w, and possibly q3w at maximum tolerated dose (MTD) (as determined in Part 2). Part 3 will only be conducted if the risk/benefit assessment, as evaluated by the Sponsor and the investigators, is in favor of the participants. Participants will be treated until disease progression, unacceptable toxicity or withdrawal from treatment for other reasons or death for a maximum duration of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed advanced and/or metastatic solid tumor, with at least one tumor lesion of non-critical location accessible to biopsy who have progressed on the standard of care therapy
* Locally confirmed CEA expression in tumor tissue (more than [>] 20 percent (%) of tumor cells staining with at least moderate intensity) or centrally confirmed CEA expression if no archival tumor tissue and fresh biopsy is collected
* Radiologically measurable and clinically evaluable disease
* Life expectancy of greater than or equal to (>/=) 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* All acute toxic effects of any prior radiotherapy, chemotherapy or surgical procedure must have resolved to Grade </=1, except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate hematological, liver, and renal function
* Negative serum pregnancy test within 7 days prior to study treatment in premenopausal women and women </=2 years after menopause
* Participants with Gilbert's syndrome will be eligible for the study. A diagnosis of Gilbert's syndrome will be based on the exclusion of other diseases based on the following criteria: (i) unconjugated hyperbilirubinemia noted on several occasions; (ii) no evidence of hemolysis (normal hemoglobin, reticulocyte count, and Lactate dehydrogenase); (iii) normal liver function tests; (iv) absence of other diseases associated with unconjugated hyperbilirubinemia

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases unless they have been previously treated, are asymptomatic and have had no requirement for steroids or enzyme inducing anticonvulsants in the last 14 days before screening
* Participants with an active second malignancy (other than non-melanoma skin cancer, or cervical carcinoma in situ). Participants who have a history of malignancy are not considered to have an active malignancy if they have completed therapy and are considered by their treating physician to be at less than (<) 30% risk for relapse
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders and known autoimmune diseases
* Uncontrolled hypertension (systolic >150 millimeter of mercury [mmHg] and/or diastolic >100 mmHg), unstable angina, congestive heart failure (CHF) of any New York Heart Association (NYHA) classification, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months of enrollment
* Active or uncontrolled infections
* Known infection with human immunodeficiency virus (HIV), seropositive status
* Positive test results for chronic hepatitis B infection (defined as positive Hepatitis B surface antigen [HBsAg] serology and/or HBcAb status)
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Pregnant or breast-feeding women
* Known hypersensitivity to any of the components of RO6895882
* Concurrent therapy with any other investigational drug
* Regular immunosuppressive therapy (that is, for organ transplantation, chronic rheumatologic disease)
* Chronic use of steroids (including inhaled) will not be allowed. Concurrent high doses of systemic corticosteroids. High dose is considered as >20 mg of dexamethasone a day (or equivalent) for >7 consecutive days
* Radiotherapy within the last 4 weeks before start of study drug treatment with the exception of limited field palliative radiotherapy for bone pain relief

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Part 2: Percentage of Participants With Dose-Limiting Toxicity (DLT) | Part 2: within 21 days after the highest dose administration
Part 2: MTD of RO6895882 | Part 2: within 21 days after the highest dose administration
Percentage of Participants With Adverse Events | Day 1 up to 28 days after last dose of study drug (up to approximately 25 months)
Percentage of Participants With Anti-drug Antibodies (ADAs) Against RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hour [Hr] 0). Part 2/3: qw schedule (1 cycle = 1 week): Predose in Cycle 1, 4, 5, 6, thereafter every 2 months; Part 2/3: q2w schedule (1 cycle = 2 weeks): Predose in Cycle 1, 4, 6, thereafter every 8 weeks. Part 2/3: q3w schedule (1 cycle = 3 weeks): Predose in Cycle 1, 2, 3, 4, 6, thereafter every 9 weeks. Additionally at treatment discontinuation or at 28-days after last dose (up to approximately 25 months)
Area Under the Serum Concentration-Time Curve (AUC) of RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Predose (Hr 0), 1 hr post start of infusion (SoI), at end of infusion (EoI), 2, 4, 24, 72, 96, 216 hrs post Day 1 dose. Part 2/3: qw schedule (1 cycle = 1 week): Predose, 1 hr post SoI, at EoI, 2, 4 hrs after EoI, 24, 72, 96 hrs postdose in Cycle 1, 5 (include 120 hrs postdose); Predose, 24, 96 hrs postdose in Cycle 2, 3, 4; Predose in any later cycle. Part 2/3: q2w schedule (1 cycle = 2 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 1, 4 (exclude 312 hrs postdose); Predose, 24, 96, 168 hrs postdose in Cycle 2; Predose in all later cycles. Part 2/3: q3w schedule (1 cycle = 3 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312, 480 hrs postdose in Cycle 1; Predose, 24, 96, 312 hrs postdose in Cycle 2; Predose, at EoI, 1, 2, 4 hrs post EoI, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 3; Predose, 24, 72, 120, 312 hrs postdose in Cycle 4; Predose in all later cycles. Maximum infusion length = 2 hrs.
Minimum Observed Serum Concentration (Cmin) of RO6895882 | Part 1/2/3: Predose (Hr 0) in all cycles (maximum up to 25 months) (cycle length = 1, 2, or 3 weeks, respectively)
Maximum Observed Serum Concentration (Cmax) of RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 216 hrs post Day 1 dose. Part 2/3: qw schedule (1 Cycle = 1 week): Predose, 1 hr post SoI, at EoI, 2, 4 hrs after EoI, 24, 72, 96 hrs postdose in Cycle 1, 5 (include 120 hrs postdose); Predose, 24, 96 hrs postdose in Cycle 2, 3, 4; Predose in any later cycle. Part 2/3: q2w schedule (1 Cycle = 2 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 1, 4 (exclude 312 hrs postdose); Predose, 24, 96, 168 hrs postdose in Cycle 2; Predose in all later cycles. Part 2/3: q3w schedule (1 Cycle = 3 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312, 480 hrs postdose in Cycle 1; Predose, 24, 96, 312 hrs postdose in Cycle 2; Predose, at EoI, 1, 2, 4 hrs post EoI, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 3; Predose, 24, 72, 120, 312 hrs postdose in Cycle 4; Predose in all later cycles. Maximum infusion length = 2 hrs.
Clearance (CL) of RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 216 hrs post Day 1 dose. Part 2/3: qw schedule (1 Cycle = 1 week): Predose, 1 hr post SoI, at EoI, 2, 4 hrs after EoI, 24, 72, 96 hrs postdose in Cycle 1, 5 (include 120 hrs postdose); Predose, 24, 96 hrs postdose in Cycle 2, 3, 4; Predose in any later cycle. Part 2/3: q2w schedule (1 Cycle = 2 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 1, 4 (exclude 312 hrs postdose); Predose, 24, 96, 168 hrs postdose in Cycle 2; Predose in all later cycles. Part 2/3: q3w schedule (1 Cycle = 3 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312, 480 hrs postdose in Cycle 1; Predose, 24, 96, 312 hrs postdose in Cycle 2; Predose, at EoI, 1, 2, 4 hrs post EoI, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 3; Predose, 24, 72, 120, 312 hrs postdose in Cycle 4; Predose in all later cycles. Maximum infusion length = 2 hrs.
Volume of Distribution at Steady State (Vss) of RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 216 hrs post Day 1 dose. Part 2/3: qw schedule (1 Cycle = 1 week): Predose, 1 hr post SoI, at EoI, 2, 4 hrs after EoI, 24, 72, 96 hrs postdose in Cycle 1, 5 (include 120 hrs postdose); Predose, 24, 96 hrs postdose in Cycle 2, 3, 4; Predose in any later cycle. Part 2/3: q2w schedule (1 Cycle = 2 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 1, 4 (exclude 312 hrs postdose); Predose, 24, 96, 168 hrs postdose in Cycle 2; Predose in all later cycles. Part 2/3: q3w schedule (1 Cycle = 3 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312, 480 hrs postdose in Cycle 1; Predose, 24, 96, 312 hrs postdose in Cycle 2; Predose, at EoI, 1, 2, 4 hrs post EoI, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 3; Predose, 24, 72, 120, 312 hrs postdose in Cycle 4; Predose in all later cycles. Maximum infusion length = 2 hrs.
Half-life (t1/2) of RO6895882 | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 216 hrs post Day 1 dose. Part 2/3: qw schedule (1 Cycle = 1 week): Predose, 1 hr post SoI, at EoI, 2, 4 hrs after EoI, 24, 72, 96 hrs postdose in Cycle 1, 5 (include 120 hrs postdose); Predose, 24, 96 hrs postdose in Cycle 2, 3, 4; Predose in any later cycle. Part 2/3: q2w schedule (1 Cycle = 2 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 1, 4 (exclude 312 hrs postdose); Predose, 24, 96, 168 hrs postdose in Cycle 2; Predose in all later cycles. Part 2/3: q3w schedule (1 Cycle = 3 weeks): Predose, 1 hr post SoI, at EoI, 2, 4, 24, 72, 96, 120, 168, 312, 480 hrs postdose in Cycle 1; Predose, 24, 96, 312 hrs postdose in Cycle 2; Predose, at EoI, 1, 2, 4 hrs post EoI, 24, 72, 96, 120, 168, 312 hrs postdose in Cycle 3; Predose, 24, 72, 120, 312 hrs postdose in Cycle 4; Predose in all later cycles. Maximum infusion length = 2 hrs.

SECONDARY OUTCOMES:
Count of Cluster of Differentiation (CD) 4+ Cells Analyzed by Flow Cytometry | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), at EoI, Day (D) 2. Part 2/3: qw schedule (1 cycle = 1 week): Cycle (C) 1: Predose, at EoI, D2, D5; C2: Predose, at EoI, D2; C3: Predose, at EoI; C4: Predose. Part 2/3: q2w schedule (1 cycle = 2 weeks): C1, C4: Predose, at EoI, D2, D5, C2: Predose, at EoI, D2; C3: Predose, at EoI. Part 2/3: q3w schedule (1 cycle = 3 weeks): C1: Predose, at EoI, Day 2, 5, 14; C3: Predose, at EoI, Day 2, 5; C2, C4: Predose, at EoI, Day 2. Maximum infusion length = 2 hrs.
Count of CD8+ Cells Analyzed by Flow Cytometry | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), at EoI, Day (D) 2. Part 2/3: qw schedule (1 cycle = 1 week): Cycle (C) 1: Predose, at EoI, D2, D5; C2: Predose, at EoI, D2; C3: Predose, at EoI; C4: Predose. Part 2/3: q2w schedule (1 cycle = 2 weeks): C1, C4: Predose, at EoI, D2, D5, C2: Predose, at EoI, D2; C3: Predose, at EoI. Part 2/3: q3w schedule (1 cycle = 3 weeks): C1: Predose, at EoI, Day 2, 5, 14; C3: Predose, at EoI, Day 2, 5; C2, C4: Predose, at EoI, Day 2. Maximum infusion length = 2 hrs.
Count of B Lymphocyte Cells Analyzed by Flow Cytometry | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), at EoI, Day (D) 2. Part 2/3: qw schedule (1 cycle = 1 week): Cycle (C) 1: Predose, at EoI, D2, D5; C2: Predose, at EoI, D2; C3: Predose, at EoI; C4: Predose. Part 2/3: q2w schedule (1 cycle = 2 weeks): C1, C4: Predose, at EoI, D2, D5, C2: Predose, at EoI, D2; C3: Predose, at EoI. Part 2/3: q3w schedule (1 cycle = 3 weeks): C1: Predose, at EoI, Day 2, 5, 14; C3: Predose, at EoI, Day 2, 5; C2, C4: Predose, at EoI, Day 2. Maximum infusion length = 2 hrs
Count of Natural Killer (NK) Cells Analyzed by Flow Cytometry | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), at EoI, Day (D) 2. Part 2/3: qw schedule (1 cycle = 1 week): Cycle (C) 1: Predose, at EoI, D2, D5; C2: Predose, at EoI, D2; C3: Predose, at EoI; C4: Predose. Part 2/3: q2w schedule (1 cycle = 2 weeks): C1, C4: Predose, at EoI, D2, D5, C2: Predose, at EoI, D2; C3: Predose, at EoI. Part 2/3: q3w schedule (1 cycle = 3 weeks): C1: Predose, at EoI, Day 2, 5, 14; C3: Predose, at EoI, Day 2, 5; C2, C4: Predose, at EoI, Day 2. Maximum infusion length = 2 hrs
Count of Monocytes Cells Analyzed by Flow Cytometry | Baseline up to 28-days after last dose (up to approximately 25 months) (please see outcome measure description for detailed time frame)
  Part 1: Predose (Hr 0), at EoI, Day (D) 2. Part 2/3: qw schedule (1 cycle = 1 week): Cycle (C) 1: Predose, at EoI, D2, D5; C2: Predose, at EoI, D2; C3: Predose, at EoI; C4: Predose. Part 2/3: q2w schedule (1 cycle = 2 weeks): C1, C4: Predose, at EoI, D2, D5, C2: Predose, at EoI, D2; C3: Predose, at EoI. Part 2/3: q3w schedule (1 cycle = 3 weeks): C1: Predose, at EoI, Day 2, 5, 14; C3: Predose, at EoI, Day 2, 5; C2, C4: Predose, at EoI, Day 2. Maximum infusion length = 2 hrs.
Percentage of Participants With Objective Response Assessed According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v 1.1) | From Screening until disease progression or death (up to approximately 25 months)
Percentage of Participants With Stable Disease Assessed According to RECIST v 1.1 | From Screening until disease progression or death (up to approximately 25 months)
Percentage of Participants With Disease Control Assessed According to RECIST v 1.1 | From Screening until disease progression or death (up to approximately 25 months)
Progression-Free Survival Assessed According to RECIST v 1.1 | From Screening until disease progression or death (up to approximately 25 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Rigshospitalet, Onkologisk Klinik, København Ø, Denmark
- Helsinki University Central Hospital; Dept of Oncology, Helsinki, Finland
- Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif, France
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
- Spain (2):
  - Clinica Universitaria de Navarra; Servicio de oncología, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
- CHUV; Departement d'Oncologie, Lausanne, Switzerland
- Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Melero I, Steeghs N, Lassen U, Homicsko K, Tabernero J, Canamero M, Roller A, Duarte J, Rossmann E, Babitzki G, Grabole N, Watson C, Habigt C, Evers S, Dejardin D, Teichgraber V, Charo J. Biomarkers of activity from a phase I study of cergutuzumab amunaleukin in patients with advanced solid tumors. J Immunother Cancer. 2026 Jan 16;14(1):e012885. doi: 10.1136/jitc-2025-012885. PMID 41545306